CLINICAL TRIAL: NCT06302634
Title: Hospital-based Cardio-Oncology Rehabilitation Care Process for Cardiovascular Health in Cancer Patients
Brief Title: Cardio-Oncology Rehabilitation Care Process
Acronym: ReCO
Status: Recruiting | Type: Observational
Sponsor: Hospital Clinico Universitario de Santiago (Other)
Responsible Party: Principal Investigator, Carlos Peña Gil, Head of Cardiac Rehabilitation Unit, Hospital Clinico Universitario de Santiago
Other Study IDs: ReCO; 2022/137 (Other: Comité de Ética de la Investigación de Santiago-Lugo)
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Cardio-Oncology; Rehabilitation; Cardiovascular Diseases; Exercise
Keywords: cardio-oncology rehabilitation; cardiovascular prevention; exercise; cancer
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Center-Based Cardio-Oncology Rehabilitation (CBCORe): Therapeutic exercise program supervised by a physiotherapist. 2 days/week, duration 1h, in the Cardiac Rehabilitation ward.
  Interventions: Other: Exercise-based cardio-oncology rehabilitation
- Home-Based Cardio-Oncology Rehabilitation (HBCORe): Recommendation of physical exercise and motivational interview through telephone follow-up every 2 weeks by the physiotherapist.
  Interventions: Other: Exercise-based cardio-oncology rehabilitation

INTERVENTIONS:
Other: Exercise-based cardio-oncology rehabilitation — Within the multidisciplinary approach of cardio-oncology rehabilitation, the exercise program will include recommendation and supervision of strength, aerobic and mobility exercises.

SUMMARY:
The objective of this observational study is to assess the outcomes of a hospital-based Cardio-Oncology Rehabilitation (CORe) program focused on exercise in cancer patients undergoing cardiotoxic treatment. This evaluation will be conducted by analyzing disease-related health indicators, functional capacity, and quality of life. Patients at risk of cardiotoxicity attending the Cardio-Onco-Hematology Unit will be offered the exercise program, which includes two modalities: in-person (center-based) and remote (home-based) options. The assignment to either modality is non randomized, based on the functional assessment conducted in the Rehabilitation Unit and the agreement between healthcare professional and patient. All participants will perform a 3-month supervised exercise intervention. There are 3 time points for assessment: at baseline (T0), 3-month after the exercise program (T1) and follow-up at 9 months from baseline (T2).

DETAILED DESCRIPTION:
Advancements in pharmacological cancer treatment have significantly improved prognosis and increased survival rates. However, the chronicity of treatment-related side effects or associated comorbidities may be exacerbated. Various chemotherapy treatments are associated with the potential development of cardiovascular diseases, such as cardiotoxicity, which stands as a main cause of death among women with early-stage breast cancer. Additionally, other side effects, such as fatigue, loss of muscle mass, insomnia, lymphedema, and cognitive impairments, can markedly decline the quality of life of these patients.

The comprehensive care of oncology patients should extend beyond curative interventions like surgery, radiotherapy, or chemotherapy. It must encompass other aspects, such as psychological support, social support and therapeutic exercise programs to enhance the overall treatment experience and improve the quality of life. Exercise has proven to reduce mortality, morbidity, and the risk of recurrence, improving treatment tolerance and reducing interruptions, thereby promoting adherence. Supervised exercise programs are increasingly recognized as a low-cost and a side-effect-free "polypill". However, they have not yet been integrated into the standard care of patients with cancer.

The inherited experience from multimodal Cardiac Rehabilitation (CR) programs with a comprehensive assessment and a multifaceted intervention with exercise programs as a central component; could be extended to cancer patients, resulting in a CORe program (ReCO in Spanish) by utilizing available CR programs in all healthcare areas.

The proposed CORe care process is grounded in the prior experience with the ONCORE trial (Clinicaltrials.gov: NCT03964142), which has helped in the implementation of new, structured, and controlled healthcare service, ensuring higher quality, safety, and efficiency in healthcare.

The implementation of the CORe program will take place at the University Hospital Complex of Santiago de Compostela (CHUS), under the coordination of the Cardiology, Oncology, and Rehabilitation services. The management of participants data and the establishment of indicators should facilitate the monitoring of the process and the evaluation of the results of clinical interventions.

The goal of this project is to assess the outcomes of a CORe care process through the analysis of health-related indicators, functional capacity, and the quality of life of breast cancer participants attending the Cardio-Oncology Unit.

ELIGIBILITY:
Inclusion Criteria:

* High risk of cancer treatment-related cardiotoxicity
* Possibility of completing a cardio-onco rehabilitation program (centre-based or home-based) and programmed visits.
* Providing written informed consent.

Exclusion Criteria:

* Patients with physical or mental limitation to carry out an exercise program.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with breast cancer at high risk of developing cardiotoxicity
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2027-06-22 (Estimated); Study Completion 2027-06-22 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricular systolic function quantified by left ventricular ejection fraction and global longitudinal strain by transthoracic echocardiography | Baseline (T0); 3 months after completing the exercise program (T1); follow-up at 9 months from baseline (T2); every year after study completion up to a maximum of 5 years
  Fall of 10 absolute percentage points of left ventricular ejection fraction from baseline or with final value below 53% or global longitudinal strain fall >15% with respect to baseline
Increased cardiac biomarkers (Troponin I and BNP/NT-proBNP) | Baseline (T0); 3 months after completing the exercise program (T1); follow-up at 9 months from baseline (T2); every year after study completion up to a maximum of 5 years
  cTnI/T>percentil 99, BNP≥35 pg/mL, NT-proBNP≥125 pg/mL
Decrease in functional capacity assessed by estimated VO2peak | Baseline (T0); 3 months after completing the exercise program (T1); follow-up at 9 months from baseline (T2)
  To estimate VO2peak, the ONCORE equation developed in the following article is used: Díaz-Balboa, E., González-Salvado, V., Rodríguez-Romero, B. et al. Thirty-second sit-to-stand test as an alternative for estimating peak oxygen uptake and 6-min walking distance in women with breast cancer: a cross-sectional study. Support Care Cancer 30, 8251-8260 (2022). https://doi.org/10.1007/s00520-022-07268-z
Change in cardiovascular risk profile as assessed by the presence or absence of classic cardiovascular risk factors. | Baseline (T0); 3 months after completing the exercise program (T1); follow-up at 9 months from baseline (T2); every year after study completion up to a maximum of 5 years
  Dyslipidemia, Diabetes mellitus, Arterial Hypertension, Smoking status
Changes in fasting blood glucose | Baseline (T0); 3 months after completing the exercise program (T1); follow-up at 9 months from baseline (T2); every year after study completion up to a maximum of 5 years
  Value of fasting blood glucose (mg/dL) in blood tests
Changes in total low-density lipoprotein (LDL) and total cholesterol (TC) levels | Baseline (T0); 3 months after completing the exercise program (T1); follow-up at 9 months from baseline (T2); every year after study completion up to a maximum of 5 years
  Value of LDL >160 mg/dL or CT> 200 mg/dL in blood tests
Change in haemoglobin | Baseline (T0); 3 months after completing the exercise program (T1); follow-up at 9 months from baseline (T2); every year after study completion up to a maximum of 5 years
  Value of haemoglobin (g/dL) in blood tests
Significant cardiovascular and non-cardiovascular adverse effects during treatment. | Date of the event throughout the study.
  number of participants with significant cardiovascular and non-cardiovascular adverse effects throughout the study, threatening life, requiring admission, prolonging hospitalization, being clinically relevant or causing chemotherapy interruptions.

SECONDARY OUTCOMES:
Change in health-related quality of life assessed by the Functional Assessment of Cancer Therapy - Breast plus Arm Morbidity (FACT-B+4) questionnaire. | Baseline (T0); 3 months after completing the exercise program (T1); follow-up at 9 months from baseline (T2)
  Score achieved in the Functional Assessment of Cancer Therapy - Breast plus Arm Morbidity (FACT-B+4) questionnaire, a specific validated scale to assess quality of life of women with breast cancer. It comprises 27 items within 5 areas of assessment: physical well-being (7 items), social and family environment (7 items), emotional well-being (7 items), functional well-being (6 items) and worries related to the diagnosis and treatment of the disease (9 items). Each item is scored by means of a Likert scale from 0 to 5, with higher scores representing better results. The total score is obtained by adding the scores for each item, and ranges from a minimum of 0 (worst possible result) to a maximum of 146 (best possible result).
Change in localized lower limb functional capacity assessed by number of repetitions performed within 30 seconds in the sit-to-stand test. | Baseline (T0); 3 months after completing the exercise program (T1); follow-up at 9 months from baseline (T2)
  Number of repetitions in the sit-to-stand test within 30 seconds.
Change in lower limb strength measured by squat dynamometry (kg). | Baseline (T0); 3 months after completing the exercise program (T1); follow-up at 9 months from baseline (T2)
  Kilograms by dynamometry.
Change in biceps strength by dynamometry (kg). | Baseline (T0); 3 months after completing the exercise program (T1); follow-up at 9 months from baseline (T2)
  Kilograms by dynamometry.
Change in perimeter (cm) of the right thigh 5cm above the upper edge of the patella | Baseline (T0); 3 months after completing the exercise program (T1); follow-up at 9 months from baseline (T2)
  Thigh perimeter measured with a tape measure in cm.
Changes in peak expiratory flow | Baseline (T0); 3 months after completing the exercise program (T1); follow-up at 9 months from baseline (T2)
  The peak expiratory flow in units of liters per minute (L/min), measured with a peak flow meter.
Change in upper limb strength measured by dynamometry (kg). | Baseline (T0); 3 months after completing the exercise program (T1); follow-up at 9 months from baseline (T2)
  Grip strength (both right and left side) and bilateral biceps strength in kilograms by dynamometry.
Change in anthropometric parameters: weight in kg. | Baseline (T0); 3 months after completing the exercise program (T1); follow-up at 9 months from baseline (T2)
  Weight measured in kg.
Change in anthropometric parameters: Body mass index (BMI) in kg/m^2 | Baseline (T0); 3 months after completing the exercise program (T1); follow-up at 9 months from baseline (T2)
  Weight and height will be combined to report BMI in kg/m^2
Change in anthropometric parameters: abdominal circumference in cm. | Baseline (T0); 3 months after completing the exercise program (T1); follow-up at 9 months from baseline (T2)
  Abdominal perimeter measured with a tape measure in cm.
Change in resting heart rate measured by pulse oximetry (beats per min). | Baseline (T0); 3 months after completing the exercise program (T1); follow-up at 9 months from baseline (T2)
  Resting heart rate by pulse oximetry (beats per min).
Change in resting blood pressure (mmHg) measured by a blood pressure monitor. | Baseline (T0); 3 months after completing the exercise program (T1); follow-up at 9 months from baseline (T2)
  Resting blood pressure by a blood pressure monitor in mmHg.
Change in physical activity assessed by the score in the Godin Leisure Test Exercise Questionnaire (GLTEQ). | Baseline (T0); 3 months after completing the exercise program (T1); follow-up at 9 months from baseline (T2).
  Score achieved in the Godin Leisure Test Exercise Questionnaire (GLTEQ) for quantification of physical activity. Activities are classified into three subgroups: "strenuous," "moderate," and "light." The scores corresponding to the energy expenditure (metabolic equivalent (MET)) are obtained by multiplying activities performed for more than 15 min in a week with their coefficients. The numbers represent the MET intensity values (strenuous/ exhausting exercises: 9 METs, moderate exercises: 5 METs, and light exercises: 3 METs).The increasing scores are associated with the increasing number of exercise behaviors, providing references about the contribution of physical activity to health: the activity score of 24 units and more as active (substantial benefits); the activity score of 14-23 units as moderately active (some benefits); and the activity score of 13 units and less as inactive (less substantial or low benefits).
Change in cardiovascular treatment by its presence or absence. | Baseline (T0); 3 months after completing the exercise program (T1); follow-up at 9 months from baseline (T2).
  ACE Inhibitor/ARB II; Beta-blocker; Statins; Ezetimibe

OTHER OUTCOMES:
Adherence and compliance to cardiac rehabilitation program (CBCORe) assessed by number of training sessions attended/number of sessions planned. | At the end of the cardiac rehabilitation program (3 months duration).
  Number of training sessions attended / number of sessions planned.
Compliance to home-based cardiac rehabilitation program (HBCORe) assessed by the total number of telephone calls during the Physiotherapy follow-up and the total time of telephone calls. | At the end of the cardiac rehabilitation program (3 months duration).
  Number of telephone calls attended / number of telephone calls planned.
Security of the cardiac rehabilitation program assessed by number of adverse events during training (CBCORe). | At the end of the cardiac rehabilitation program (3 months duration).
  Adverse events during training.
Satisfaction with the CORe program | At the end of the cardiac rehabilitation program (3 months duration).
  Global satisfaction is scored from 0 (no benefit) to 10 (highest benefit); and evaluated with an open-ended question, how do you expect to benefit from participating in the program?
Follow-up of the exercise performed after participation in the CORe program | At follow-up at 9 months from baseline (T2).
  Question (yes/no): do you continue exercising? supervized? if supervized, is it individualized by a physiotherapist? individualized by a personal trainer? recommendations from a technician in a gym? or city council group activities?
Presence or absence of lymphoedema. | Baseline (T0); 3 months after completing the exercise program (T1); follow-up at 9 months from baseline (T2).
  It is considered 2 cm difference between upper limbs. Measurement is performed at the base of the 3rd finger, hand, wrist, 10 cm above the wrist, elbow, 10 cm above the elbow and axilla.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Peña-Gil, MD, PhD, Study Director — Hospital Clinico Universitario de Santiago; Violeta González-Salvado, MD, PhD, Study Chair — Hospital Clinico Universitario de Santiago
Locations (1):
- Hospital Clínico Universitario de Santiago, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Shared in the institutional repository of SERGAS (RUNA), upon request